CLINICAL TRIAL: NCT07326306
Title: Dialysis Patients' Perspectives: A Study of the Q Methodology
Status: Recruiting | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Yavuz Uren, Principal Inverstigator, Yuzuncu Yil University
Other Study IDs: PD-HD Q2
Record Dates: First submitted 2025-12-22; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Dialysis Patients
Keywords: Q methodology; Peritoneal dialysis; Hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was conducted to systematically examine the subjective experiences and perspectives of dialysis patients regarding their treatment modalities.

DETAILED DESCRIPTION:
In this study, Q methodology was used to systematically examine dialysis patients' subjective experiences and perspectives regarding treatment modalities. Q methodology is a research method that combines qualitative and quantitative paradigms, requiring participants to rank statements expressing their thoughts on a specific topic according to their own perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years of age,
* Being able to read and write,
* Not having vision or hearing problems,
* Voluntary participation in our study,
* Being conscious,
* Being a patient with end-stage renal failure,
* Not having communication problems

Exclusion Criteria:

• Wishing to withdraw from the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The hospital where the study will be conducted has a total of 13 adult peritoneal dialysis patients and 70 adult hemodialysis patients who regularly receive dialysis treatment and attend follow-up appointments. The aim is to study the entire peritoneal dialysis patient population. For hemodialysis patients, a similar number of patients (n=13) to the peritoneal dialysis patients will be selected using a simple randomization method, and these patients will be included in the study.
Sampling Method: Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Perception of dialysis treatment | up to 6 months
  Hemodialysis patients were asked to rank 24 Q items, developed based on literature review and clinical experience, on a scale from -3 (strongly disagree) to +3 (strongly agree) according to a normal distribution model.

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Uren, PhD, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Sbu. Van Training and Research Hospital, Van, Turkey (Türkiye)